CLINICAL TRIAL: NCT01521806
Title: Effects of Dieatry Fiber on Insulin Sensitivity in Pre- and Post-menopausal Women
Brief Title: Effects of Dietary Fiber on Insulin Sensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HM001
Record Dates: First submitted 2012-01-20; First posted 2012-01-31 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Focus of the Study is Insulin Sensitivity
Keywords: insulin sensitivity; resistant starch
MeSH Terms: conditions — Insulin Resistance | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (Experimental): 15 g of fiber per day will be added to snack foods
  Interventions: Dietary Supplement: Dietary Fiber
- High dose (Experimental): 30 g of fiber per day will be added to snack foods
  Interventions: Dietary Supplement: Dietary Fiber
- No fiber (Placebo Comparator): Snack foods without fiber will be given
  Interventions: Dietary Supplement: Dietary Fiber

INTERVENTIONS:
Dietary Supplement: Dietary Fiber — Dietary fiber will be added to snack foods

SUMMARY:
This study will examine the effects of a dietary fiber on insulin sensitivity in overweight and obese women. The fiber will be added to snack foods and women will consume the foods for four weeks. In one four-week period, 15 g of fiber will be added, and 30 g will added in another period. In a third period, no fiber will be added to the snack foods. Insulin senstivity will be measured at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Impaired fasting glucose
* Overweight and obese

Exclusion Criteria:

* Diabetes, Presence of chronic diseases

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 5-hr test, performed 3 times within a 20-week period
  A frequently sampled intravenous blood glucose tolerance test will be performed.

SECONDARY OUTCOMES:
Mitocondrial function | 3 times, with a 20-week period
  A muscle biospy will be taken to assess mitochondrial function
Meal tolerance test | 3 times, within a 20-week period
  A high-fat meal will be given and blood will be drawn over a three-hr period

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gower, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Clinical Research Unit, Birmingham, Alabama, United States

REFERENCES:
- See also: clinical center — http://www.uab.edu/cores/clinical-research-unit-cru